CLINICAL TRIAL: NCT00927134
Title: Phase I/II Gene Therapy Study for X-linked Chronic Granulomatous Disease in Children
Brief Title: Gene Therapy for X-linked Chronic Granulomatous Disease (CGD) in Children
Acronym: XCGDinChildren
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Goethe University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PedsZürich_GT05
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic Granulomatous Disease in children (=or< 18 years)
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: retroviral SF71-gp91phox transduced CD34+ cells — autologous ex-vivo transduced (SF71-gp91phox)CD34+ cells

SUMMARY:
The aim of the study is to evaluate the side effects and risks after infusion of retroviral gene corrected autologous CD34+ cells of the peripheral blood of chemotherapy conditioned (busulphan) children with chronic granulomatous disease (CGD). Also gene corrected and functional active granulocytes in the peripheral blood and the engraftment in the bone marrow of the patients will be monitored an documented.

ELIGIBILITY:
Inclusion Criteria:

* x-linked Chronic Granulomatous Disease
* history of life-threatening severe infections
* no HLA-matched related or unrelated donor
* therapy resistent life threatening infections/organ dysfunction
* no other treatment options e.g. HSCT

Exclusion Criteria:

* > 18 years of age
* HIV infection
* life expectancy > 2 years
* infections treatable by conventional therapy (antibiotics, antimycotics, allogeneic granulocytes)

Ages: 1 Year to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2004-06; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
eradication of pre-existing therapy refractory bacterial and/or fungal infections | 6 months

SECONDARY OUTCOMES:
Reconstitution of ROS production by peripheral blood cells | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Seger, Prof Dr med, Principal Investigator — University Children's Hospital, Zurich; Janine Reichenbach, PD Dr med, Study Chair — University Children's Hospital, Zurich; Ulrich Siler, Dr rer nat, Study Chair — University Children's Hospital, Zurich; Manuel Grez, Dr rer nat, Study Chair — Georg Speyer Research Institute, Frankfurt a.M.
Locations (1):
- University Children's Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Ott MG, Schmidt M, Schwarzwaelder K, Stein S, Siler U, Koehl U, Glimm H, Kuhlcke K, Schilz A, Kunkel H, Naundorf S, Brinkmann A, Deichmann A, Fischer M, Ball C, Pilz I, Dunbar C, Du Y, Jenkins NA, Copeland NG, Luthi U, Hassan M, Thrasher AJ, Hoelzer D, von Kalle C, Seger R, Grez M. Correction of X-linked chronic granulomatous disease by gene therapy, augmented by insertional activation of MDS1-EVI1, PRDM16 or SETBP1. Nat Med. 2006 Apr;12(4):401-9. doi: 10.1038/nm1393. Epub 2006 Apr 2. PMID 16582916